CLINICAL TRIAL: NCT02236325
Title: Brief Skills Training Intervention for Suicidal Individuals
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Erin Ward-Ciesielski, Graduate student, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 40846-G
Record Dates: First submitted 2014-08-27; First posted 2014-09-10 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Suicide
MeSH Terms: conditions — Suicide | interventions — Relaxation Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DBT Brief Suicide Intervention (Experimental)
  Interventions: Behavioral: DBT Brief Suicide Intervention
- Relaxation Training (Active Comparator)
  Interventions: Behavioral: Relaxation Training

INTERVENTIONS:
Behavioral: DBT Brief Suicide Intervention — Participants assigned to the DBT Brief Suicide Intervention are presented with a selection of coping strategies selected from the Dialectical Behavior Therapy (DBT) skills training curriculum. The strategies are 1) mindfulness, 2) mindfulness of current emotions, 3) opposite-to-emotion action, 4) distraction, and 5) changing your body chemistry.
  Arms: DBT Brief Suicide Intervention
Behavioral: Relaxation Training — Participants assigned to the Relaxation Training condition receive instruction in a sensory awareness practice and are guided through the practice by the therapist.
  Arms: Relaxation Training

SUMMARY:
A significant percentage of individuals who die by suicide do not seek mental health services in the time preceding their death. This population is underserved and it is unclear what barriers keep them from seeking treatment. In order to begin a line of research aimed at addressing this high-risk population, this proposal rests on the hypothesis that suicidal individuals who do not seek treatment prior to attempting suicide experience the same psychopathological difficulties as suicidal individuals who do seek treatment - namely, severe emotion dysregulation. However, these non-treatment-seeker s will likely require more creative recruitment strategies and briefer interventions than treatment-seeking individuals. As such, this application proposes to use wide-reaching recruitment efforts throughout the community to locate and enroll individuals who are suicidal but not seeking treatment. Further, there is a paucity of empirical support for interventions targeting suicidal individuals. Dialectical Behavior Therapy (DBT) is one of the few treatments that have been demonstrated to be effective with a suicidal population and is the only treatment whose effectiveness has been replicated. Previous research has suggested that an abbreviated version of the skills that are taught in DBT skills training have effectively reduced emotion dysregulation (i.e., depression and anxiety) in problem drinkers and the format of the proposed intervention is derived from this evidence-based emotion dysregulation intervention. As such, the proposed research is a randomized, controlled pilot trial of a very brief, one-time, skills-based intervention targeting difficulties in emotion regulation and distress tolerance.

This research aims to evaluate the safety of the intervention, the feasibility of the research methods (including the appropriateness of the relaxation training control condition), and to preliminarily estimate the immediate (one week) and long-term (one and three month) changes resulting from the DBT Brief Skills Intervention (DBT-BSI) relative to a relaxation training control on the primary outcomes of suicide ideation and emotion dysregulation as well as a number of secondary outcomes. These results will inform the design of a subsequent full-scale randomized controlled trial of the DBT-BSI.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* Suicidal ideation in the last week
* Live within commuting distance to research office
* Have not been engaged in mental health treatment in the past month
* Consent to assessment

Exclusion Criteria:

* Non-English speaking
* Significant cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2012-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Scale for Suicidal Ideation | 12-weeks of follow-up
Difficulties in Emotion Regulation Scale | 12-weeks of follow-up
DBT Ways of Coping Scale | 12-weeks of follow-up

SECONDARY OUTCOMES:
Patient Health Questionnaire - Depression Module | 12-weeks of follow-up
Beck Anxiety Inventory | 12-weeks of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Erin Ward-Ciesielski, M.S., Principal Investigator — University of Washington

REFERENCES:
- [Derived] Ward-Ciesielski EF, Jones CB, Wielgus MD, Wilks CR, Linehan MM. Single-session dialectical behavior therapy skills training versus relaxation training for non-treatment-engaged suicidal adults: a randomized controlled trial. BMC Psychol. 2016 Mar 24;4:13. doi: 10.1186/s40359-016-0117-4. PMID 27009317